CLINICAL TRIAL: NCT02454088
Title: A Single-Center Investigator-Initiated Evaluator-Bilateral-Comparison Pilot Study of Injectable Calcium Hydroxylapatite With and Without Triamcinolone Acetate for the Treatment of Volume Loss to Dorsum Areas of the Hands
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Goldman, Butterwick, Fitzpatrick and Groff (Other)
Collaborators: Merz North America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RAD-2010
Record Dates: First submitted 2015-05-13; First posted 2015-05-27 (Estimated); Last update posted 2017-03-01 (Actual); Status verified 2017-02

CONDITIONS: Volume Loss to Dorsum of Hands
Keywords: Volume; Hands; Filler; Radiesse; Calcium hydroxylapatite
MeSH Terms: interventions — Triamcinolone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Triamcinolone acetate (Active Comparator): Injection of Calcium hydroxylapatite with Triamcinolone acetate
  Interventions: Other: Calcium Hydroxylapatite and Triamcinolone acetate
- Placebo (Placebo Comparator): Injection of Calcium hydroxylapatite with a placebo
  Interventions: Device: Calcium Hydroxylapatite and Placebo

INTERVENTIONS:
Other: Calcium Hydroxylapatite and Triamcinolone acetate — Combination Therapy Triamcinolone acetate and Calcium Hydroxylapatite
  Arms: Triamcinolone acetate
Device: Calcium Hydroxylapatite and Placebo — Calcium Hydroxylapatite and Placebo
  Arms: Placebo

SUMMARY:
This will be a single-center, investigator-initiated, double-blinded, randomized, bilateral-comparison pilot study of injectable Calcium hydroxylapatite with and without Triamcinolone acetate for the treatment of volume loss to the dorsum areas of the hands.

ELIGIBILITY:
Inclusion Criteria:

1. Cutaneous and soft tissue atrophy in the dorsum of both hands, as indicated by the Merz Validated Hand Grading Scale score of 2, 3 or 4.
2. Males or females in good general health who are 22 years of age or older.
3. Must be willing to give and sign an informed consent form and photographic release form.
4. Subject is planning re-volumizing rejuvenation treatment to the dorsum area of both hands.
5. For female subjects of childbearing potential, must be willing to use an acceptable form of birth control during the entire course of the study. All systemic birth control measures must be in consistent use for at least 30 days prior to study enrollment participation.

   A female is considered of childbearing potential unless she is postmenopausal, without a uterus and/or both ovaries, or has had a bilateral tubal ligation.

   Acceptable methods of birth control are: oral contraceptives, contraceptive patches/rings/implants, Implanon®, Depo-Provera®, double-barrier methods (e.g. condoms and spermicide), abstinence and/or vasectomies of partner with a documented second acceptable method of birth control, should the subject become sexually active.
6. Negative urine pregnancy test results at the time of study entry (if applicable).
7. Must be willing to comply with study dosing and complete the entire course of the study.

Exclusion Criteria:

1. A subject with any uncontrolled systemic disease. A potential subject in whom therapy for a systemic disease is not yet stabilized will not be considered for entry into the study.
2. A Subject that is currently using systemic steroids.
3. A subject with a significant history or current evidence of a medical, psychological or other disorder that, in the investigator's opinion, would preclude enrollment into the study.
4. A subject with history of or the presence of any skin condition/disease that might interfere with the diagnosis or evaluation of study parameters (i.e., atopic dermatitis, eczema, psoriasis).
5. A subject with an active bacterial, fungal, or viral infection in the treatment area.
6. A subject with an active systemic fungal infection.
7. A subject with a prior history of an allergy to any of the products or medications being used in the study.
8. A subject planning any other cosmetic procedure to the study area during the study period, other than the treatments that will be performed by the investigator.
9. A subject with a history of previous fat transfer or injectable poly-l-lactic acid to the study area within the past five years.
10. A subject with a previous history of calcium hydroxylapatite to the treatment area within the past year.
11. A subject with a previous history of ablative laser surgery to the treatment area within the past year.
12. A female subject who is pregnant, nursing an infant or planning a pregnancy during the study.
13. Subjects with known autoimmune disease or compromised immune systems i.e. HIV, AIDS or current chemotherapy.
14. Subjects with known bleeding disorder or is receiving medication that will likely increase the risk of bleeding as the result of injection per investigator discretion.
15. Subjects with a history hypertrophic scarring.
16. Subjects with a cancerous or precancerous lesion, or unhealed wound in the treatment area.
17. Current participation or participation within 30 days prior to the start of this study in a drug or other investigational research study.

Min Age: 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-05; Primary Completion 2016-10 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Efficacy Analysis (Merz Validated Hand Grading Score) | Through day 360
  The primary analyses of efficacy will be based on the change from Baseline through Day 360 for assessment (based on the Merz Validated Hand Grading Score).

CONTACTS AND LOCATIONS:
Overall Officials: Mitchel P Goldman, MD, Principal Investigator — Cosmetic Laser Dermatology
Locations (1):
- Cosmetic Laser Dermatology, San Diego, California, United States